CLINICAL TRIAL: NCT05990972
Title: To Investigate the Efficacy and Safety of Fecal Microbiota Transplantation (FMT) in the Treatment of Antibiotic-associated Diarrhea.
Brief Title: Clinical Study of Fecal Microbiota Transplantation in the Treatment of Antibiotic-associated Diarrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Huanlong Qin, Clinical Professor, Shanghai 10th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMT-AAD
Record Dates: First submitted 2023-08-07; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Fecal Microbiota Transplantation; Antibiotic-associated Diarrhea
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FMT group (Experimental)
  Interventions: Procedure: Fecal Microbiota Transplantation

INTERVENTIONS:
Procedure: Fecal Microbiota Transplantation — Fecal Microbiota Transplantation (FMT) is a therapeutic method to transplant the microbiota from the feces of healthy people into the intestinal tract of patients. This treatment aims to improve a range of diseases associated with the gut microbiota by restoring the balance of the gut microbiota.

SUMMARY:
Antibiotic-associated diarrhea (AAD) refers to the occurrence of other unexplained diarrhea symptoms after the use of antibiotics, often combined with abdominal pain, bloating and bloody stool. Fecal Microbiota Transplantation (FMT) is a therapeutic method to transplant the microbiota from the feces of healthy people into the intestinal tract of patients. To explore the overall efficacy and safety of FMT in the treatment of AAD.

ELIGIBILITY:
Inclusion Criteria:

* occurrence of antibiotic-associated diarrhoea; no response to standard therapy; agree to receive FMT and sign informed consent; willingness to provide stool samples.

Exclusion Criteria:

* non-antibiotic-associated diarrhea; did not accept FMT or did not sign informed consent; unwillingness to provide stool samples.

Ages: 21 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Changes in defecation frequency after FMT. | Baseline and three months after treatment
Changes in gut microbiota after FMT. | Baseline and three months after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Le Wang, Principal Investigator — Intestinal Microenvironment Treatment Center of General Surgery, Shanghai Tenth People's Hospital, Tenth People's Hospital of Tongji University
Locations (1):
- Intestinal Microenvironment Treatment Center of General Surgery, Shanghai Tenth People's Hospital, Tenth People's Hospital of Tongji University, Shanghai, China